CLINICAL TRIAL: NCT00688324
Title: Biomarker Study of Acamprosate in Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Alliance for Research on Schizophrenia and Depression (Other); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Robert Buchanan, Chief, Maryland Psychiatric Research Center, Outpatient Research Program, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HP-00043248; R03AA019571 (NIH)
Record Dates: First submitted 2008-05-28; First posted 2008-06-02 (Estimated); Results first posted 2018-01-23 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: schizophrenia; schizoaffective disorder; glutamate; NMDA receptor; magnetic resonance spectroscopy; acamprosate
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Acamprosate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm (Experimental): All subjects will have baseline measures, receive acamprosate for 2 weeks, then have measures repeated.
  Interventions: Drug: Acamprosate

INTERVENTIONS:
Drug: Acamprosate — Acamprosate 333mg, ii tablets PO tid x 2 weeks
  Other Names: Campral

SUMMARY:
NMDA receptors are brain receptors that are stimulated by glutamate. Poorly functioning NMDA receptors are thought to be involved in the pathology of schizophrenia. This hypothesis is based on the observation that PCP, which blocks the NMDA receptor, produces symptoms and cognitive impairments similar to schizophrenia. Efforts to enhance the function of the NMDA receptor with glycine and D-cycloserine have met with limited success. An alternative approach would be to use the drug acamprosate.

Acamprosate, FDA-approved for maintenance of sobriety after detoxification from alcohol, seems to act through modulation of the NMDA receptor. In the lab, acamprosate has been noted to act as an antagonist when the NMDA receptors are maximally stimulated but as an agonist when NMDA receptor stimulation is minimal. This "smart drug" action makes acamprosate appealing for use in schizophrenia. If acamprosate works as a smart drug in patients, then we would predict that it would enhance the function of NMDA receptors in schizophrenia and improve cognition and the symptoms of the illness. Additionally, acamprosate seems to modulate the NMDA receptor in novel ways distinct from glycine and D-cycloserine.

We will also see if the response to acamprosate differs based on whether participants do or do not have a past history of alcohol use disorders.

DETAILED DESCRIPTION:
We propose to measure the response of symptoms and cognition in people schizophrenia given acamprosate or placebo. We hypothesize that symptoms and cognition will improve following two weeks of acamprosate. We will also use proton magnetic resonance spectroscopy (MRS) to examine the effect of acamprosate on glutamate & glutamine (Glu&Gln) brain levels in people with schizophrenia. We hypothesize that Glu&Gln concentrations in people with chronic schizophrenia will increase following two weeks of treatment with acamprosate.

The proposed study will consist of 50 individuals with chronic schizophrenia/schizoaffective disorder, 18-55 years old, from in/outpatient programs at the Maryland Psychiatric Research Center (MPRC). The dose of acamprosate will follow manufacturer recommendations with two 333mg tablets given three times per day. MRS will be acquired from areas involved in schizophrenia [dorsolateral-prefrontal cortex (DLPFC) and anterior cingulate cortex (ACC)] at baseline and week two. Symptom ratings and cognitive testing will occur at baseline and be repeated at week two.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosis of schizophrenia/schizoaffective disorder
* Age 18-55 years
* Male or female
* Any Race/ethnicity
* Participants will be analyzed separately depending on whether they do or do not have a history of an alcohol use disorder

Exclusion Criteria:

* Pregnant/nursing females or females not using adequate birth control
* Documented history of mental retardation/severe neurological disorder/head injury with loss of consciousness
* DSM-IV diagnosis of substance dependence in previous six months/abuse in the previous three months (except nicotine)
* Serious suicidal risk in the previous six months
* History of renal failure/creatinine clearance of less than 50mL/min
* Current treatment with clozapine
* Contraindication to MRI scanning.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2008-06 (Actual); Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bernard A Fischer, M.D., Principal Investigator — Food and Drug Administration (FDA)
Locations (4):
- United States (4):
  - VA Maryland Health Care System, Baltimore, Maryland
  - Keypoint Community Mental Health Centers- Dundalk, Baltimore, Maryland
  - Keypoint Community Mental Health Centers- Catonsville, Baltimore, Maryland
  - Maryland Psychiatric Research Center, Baltimore, Maryland

REFERENCES:
- See also: Maryland Psychiatric Research Center — http://www.mprc.umaryland.edu/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were 39 subjects who signed consent for the study. Three subjects were excluded prior to entering the study: two subjects refused to continue and one subject was hospitalized. Thirty six subjects entered the first phase of the study.
Period: Overall Study
Arm/Group | Single Arm
Started | 36
Completed | 28
Not Completed | 8
Not completed — Withdrawal by Subject | 2
Not completed — Physician Decision | 5
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Groups:
- Baseline Screening: All subjects will have baseline measures
Arm/Group | Baseline Screening
Number analyzed (Participants) | 36
Age, Categorical [Count of Participants; unit: Participants] — Population: Date of birth was not recorded for eight participants who gave consent for screening but did not complete the study.
  Participants
    number analyzed (Participants) | 28
    <=18 years | 0
    Between 18 and 65 years | 28
    >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Date of birth was not recorded for eight participants who gave consent for screening but did not complete the study.
  years
    number analyzed (Participants) | 28
    (all) | 44 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 34
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 20
  White | 12
  More than one race | 3
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 36
Alcohol Abuse History [Number; unit: participants]
  Present | 16
  Absent | 18
  Missing | 2

OUTCOME MEASURES:

1. Primary Outcome: Anterior Cingulate Cortex - Choline
Description: Choline brain metabolite levels between those with and without a lifetime history of prior alcohol abuse/dependence in the Anterior Cingulate Cortex (ACC) using Magnetic Resonance Spectroscopy (MRS). Metabolite concentration was calculated from the MRS signals and reported in "mM".
Time Frame: Baseline screening (Scan 1) and again after 2 weeks of Acamprosate treatment (Scan 2)
Population: Subjects entering baseline screening minus the two subjects with missing alcohol abuse history.
Measure: Mean (Standard Deviation); unit: mM
Groups:
- ETOH Abuse: Lifetime History of Alcohol Abuse/Dependence
- No ETOH Abuse: No Lifetime History of Alcohol Abuse/Dependence
Arm/Group | ETOH Abuse | No ETOH Abuse
Number analyzed (Participants) | 16 | 18
mM
  Scan 1 | 1.64 (0.20) | 1.54 (0.26)
  Scan 2: number analyzed (Participants) | 11 | 15
  Scan 2 | 1.46 (0.18) | 1.58 (0.26)
  Difference: number analyzed (Participants) | 11 | 15
  Difference | -0.10 (0.12) | 0.04 (0.19)

2. Primary Outcome: Anterior Cingulate Cortex - Creatinine
Description: Creatinine brain metabolite levels between those with and without a lifetime history of prior alcohol abuse/dependence in the Anterior Cingulate Cortex (ACC) using Magnetic Resonance Spectroscopy (MRS). Metabolite concentration was calculated from the MRS signals and reported in "mM".
Time Frame: Baseline screening (Scan 1) and again after 2 weeks of Acamprosate treatment (Scan 2)
Population: Subjects entering baseline screening minus the two subjects with missing alcohol abuse history.
Measure: Mean (Standard Deviation); unit: mM
Arm/Group | ETOH Abuse | No ETOH Abuse
Number analyzed (Participants) | 16 | 18
mM
  Scan 1 | 5.46 (0.61) | 5.12 (0.81)
  Scan 2: number analyzed (Participants) | 11 | 15
  Scan 2 | 5.09 (0.54) | 5.16 (0.74)
  Difference: number analyzed (Participants) | 11 | 18
  Difference | -0.14 (0.31) | 0.07 (0.39)

3. Primary Outcome: Anterior Cingulate Cortex - Glutamate
Description: Glutamate brain metabolite levels between those with and without a lifetime history of prior alcohol abuse/dependence in the Anterior Cingulate Cortex (ACC) using Magnetic Resonance Spectroscopy (MRS). Metabolite concentration was calculated from the MRS signals and reported in "mM".
Time Frame: Baseline screening (Scan 1) and again after 2 weeks of Acamprosate treatment (Scan 2)
Population: Subjects entering baseline screening minus the two subjects with missing alcohol abuse history.
Measure: Mean (Standard Deviation); unit: mM
Arm/Group | ETOH Abuse | No ETOH Abuse
Number analyzed (Participants) | 16 | 18
mM
  Scan 1 | 7.44 (0.65) | 6.68 (1.86)
  Scan 2: number analyzed (Participants) | 11 | 18
  Scan 2 | 7.06 (0.78) | 7.05 (2.02)
  Difference: number analyzed (Participants) | 11 | 18
  Difference | -0.25 (0.91) | 0.26 (1.28)

4. Primary Outcome: Anterior Cingulate Cortex - N-acetylaspartate
Description: N-acetylaspartate (NAA) brain metabolite levels between those with and without a lifetime history of prior alcohol abuse/dependence in the Anterior Cingulate Cortex (ACC) using Magnetic Resonance Spectroscopy (MRS). Metabolite concentration was calculated from the MRS signals and reported in "mM".
Time Frame: Baseline screening (Scan 1) and again after 2 weeks of Acamprosate treatment (Scan 2)
Population: Subjects entering baseline screening minus the two subjects with missing alcohol abuse history.
Measure: Mean (Standard Deviation); unit: mM
Arm/Group | ETOH Abuse | No ETOH Abuse
Number analyzed (Participants) | 16 | 18
mM
  Scan 1 | 6.40 (0.52) | 5.99 (1.11)
  Scan 2: number analyzed (Participants) | 11 | 15
  Scan 2 | 6.06 (0.59) | 6.14 (0.86)
  Difference: number analyzed (Participants) | 11 | 15
  Difference | -0.23 (0.35) | 0.15 (0.53)

5. Primary Outcome: Anterior Cingulate Cortex - Myo-inositol
Description: Myo-inositol brain metabolite levels between those with and without a lifetime history of prior alcohol abuse/dependence in the Anterior Cingulate Cortex (ACC) using Magnetic Resonance Spectroscopy (MRS). Metabolite concentration was calculated from the MRS signals and reported in "mM".
Time Frame: Baseline screening (Scan 1) and again after 2 weeks of Acamprosate treatment (Scan 2)
Population: Subjects entering baseline screening minus the two subjects with missing alcohol abuse history.
Measure: Mean (Standard Deviation); unit: mM
Arm/Group | ETOH Abuse | No ETOH Abuse
Number analyzed (Participants) | 16 | 18
mM
  Scan 1 | 4.34 (0.53) | 4.00 (1.34)
  Scan 2: number analyzed (Participants) | 11 | 14
  Scan 2 | 4.00 (0.67) | 4.35 (0.81)
  Difference: number analyzed (Participants) | 11 | 14
  Difference | -0.17 (0.46) | 0.20 (0.46)

6. Primary Outcome: Right Dorsal Lateral Prefrontal Cortex - Choline
Description: Choline brain metabolite levels between those with and without a lifetime history of prior alcohol abuse/dependence in the Right Dorsal Lateral Prefrontal Cortex (R DLPFC) using Magnetic Resonance Spectroscopy (MRS). Metabolite concentration was calculated from the MRS signals and reported in "mM".
Time Frame: Baseline screening (Scan 1) and again after 2 weeks of Acamprosate treatment (Scan 2)
Population: Usable scan data.
Measure: Mean (Standard Deviation); unit: mM
Arm/Group | ETOH Abuse | No ETOH Abuse
Number analyzed (Participants) | 13 | 17
mM
  Scan 1 | 1.36 (0.29) | 1.30 (0.29)
  Scan 2: number analyzed (Participants) | 8 | 15
  Scan 2 | 1.32 (0.17) | 1.71 (1.11)
  Difference: number analyzed (Participants) | 7 | 15
  Difference | 0.06 (0.16) | 0.40 (1.20)

7. Primary Outcome: Right Dorsal Lateral Prefrontal Cortex - Creatinine
Description: Creatinine brain metabolite levels between those with and without a lifetime history of prior alcohol abuse/dependence in the Right Dorsal Lateral Prefrontal Cortex (R DLPFC) using Magnetic Resonance Spectroscopy (MRS). Metabolite concentration was calculated from the MRS signals and reported in "mM".
Time Frame: Baseline screening (Scan 1) and again after 2 weeks of Acamprosate treatment (Scan 2)
Population: Usable scan data.
Measure: Mean (Standard Deviation); unit: mM
Arm/Group | ETOH Abuse | No ETOH Abuse
Number analyzed (Participants) | 15 | 17
mM
  Scan 1 | 5.51 (0.61) | 5.48 (0.92)
  Scan 2: number analyzed (Participants) | 11 | 15
  Scan 2 | 5.52 (0.51) | 5.54 (0.70)
  Difference: number analyzed (Participants) | 10 | 15
  Difference | 0.27 (0.64) | 0.11 (0.76)

8. Primary Outcome: Right Dorsal Lateral Prefrontal Cortex - Glutamate
Description: Glutamate brain metabolite levels between those with and without a lifetime history of prior alcohol abuse/dependence in the Right Dorsal Lateral Prefrontal Cortex (R DLPFC) using Magnetic Resonance Spectroscopy (MRS). Metabolite concentration was calculated from the MRS signals and reported in "mM".
Time Frame: Baseline screening (Scan 1) and again after 2 weeks of Acamprosate treatment (Scan 2)
Population: Usable scan data.
Measure: Mean (Standard Deviation); unit: mM
Arm/Group | ETOH Abuse | No ETOH Abuse
Number analyzed (Participants) | 13 | 15
mM
  Scan 1 | 6.89 (1.10) | 7.51 (2.00)
  Scan 2: number analyzed (Participants) | 11 | 13
  Scan 2 | 6.63 (1.03) | 7.15 (0.92)
  Difference: number analyzed (Participants) | 9 | 12
  Difference | -0.44 (1.52) | -0.69 (1.90)

9. Primary Outcome: Right Dorsal Lateral Prefrontal Cortex - N-acetylaspartate
Description: N-acetylaspartate (NAA) brain metabolite levels between those with and without a lifetime history of prior alcohol abuse/dependence in the Right Dorsal Lateral Prefrontal Cortex (R DLPFC) using Magnetic Resonance Spectroscopy (MRS). Metabolite concentration was calculated from the MRS signals and reported in "mM".
Time Frame: Baseline screening (Scan 1) and again after 2 weeks of Acamprosate treatment (Scan 2)
Population: Usable scan data.
Measure: Mean (Standard Deviation); unit: mM
Arm/Group | ETOH Abuse | No ETOH Abuse
Number analyzed (Participants) | 15 | 17
mM
  Scan 1 | 7.43 (0.78) | 7.65 (1.03)
  Scan 2: number analyzed (Participants) | 11 | 15
  Scan 2 | 7.65 (0.54) | 8.15 (1.24)
  Difference: number analyzed (Participants) | 10 | 15
  Difference | 0.35 (0.78) | 0.42 (0.96)

10. Primary Outcome: Right Dorsal Lateral Prefrontal Cortex - Myo-inositol
Description: Myo-inositol brain metabolite levels between those with and without a lifetime history of prior alcohol abuse/dependence in the Right Dorsal Lateral Prefrontal Cortex (R DLPFC) using Magnetic Resonance Spectroscopy (MRS). Metabolite concentration was calculated from the MRS signals and reported in "mM".
Time Frame: Baseline screening (Scan 1) and again after 2 weeks of Acamprosate treatment (Scan 2)
Population: Usable scan data.
Measure: Mean (Standard Deviation); unit: mM
Arm/Group | ETOH Abuse | No ETOH Abuse
Number analyzed (Participants) | 15 | 16
mM
  Scan 1 | 3.73 (0.72) | 3.71 (0.43)
  Scan 2: number analyzed (Participants) | 11 | 14
  Scan 2 | 3.41 (0.43) | 3.44 (0.68)
  Difference: number analyzed (Participants) | 10 | 14
  Difference | -0.17 (0.66) | -0.24 (0.76)

11. Primary Outcome: Left Dorsal Lateral Prefrontal Cortex - Choline
Description: Choline brain metabolite levels between those with and without a lifetime history of prior alcohol abuse/dependence in the Left Dorsal Lateral Prefrontal Cortex (L DLPFC) using Magnetic Resonance Spectroscopy (MRS). Metabolite concentration was calculated from the MRS signals and reported in "mM".
Time Frame: Baseline screening (Scan 1) and again after 2 weeks of Acamprosate treatment (Scan 2)
Population: Usable scan data.
Measure: Mean (Standard Deviation); unit: mM
Arm/Group | ETOH Abuse | No ETOH Abuse
Number analyzed (Participants) | 16 | 15
mM
  Scan 1 | 1.53 (0.36) | 1.53 (0.23)
  Scan 2: number analyzed (Participants) | 11 | 13
  Scan 2 | 1.57 (0.20) | 1.65 (0.21)
  Difference: number analyzed (Participants) | 10 | 13
  Difference | 0.05 (0.24) | 0.10 (0.23)

12. Primary Outcome: Left Dorsal Lateral Prefrontal Cortex - Creatinine
Description: Creatinine brain metabolite levels between those with and without a lifetime history of prior alcohol abuse/dependence in the Left Dorsal Lateral Prefrontal Cortex (L DLPFC) using Magnetic Resonance Spectroscopy (MRS). Metabolite concentration was calculated from the MRS signals and reported in "mM".
Time Frame: Baseline screening (Scan 1) and again after 2 weeks of Acamprosate treatment (Scan 2)
Population: Usable scan data.
Measure: Mean (Standard Deviation); unit: mM
Arm/Group | ETOH Abuse | No ETOH Abuse
Number analyzed (Participants) | 17 | 15
mM
  Scan 1 | 5.38 (0.84) | 5.78 (0.64)
  Scan 2: number analyzed (Participants) | 12 | 13
  Scan 2 | 5.43 (1.13) | 5.86 (0.53)
  Difference: number analyzed (Participants) | 12 | 13
  Difference | 0.15 (0.82) | 0.11 (0.55)

13. Primary Outcome: Left Dorsal Lateral Prefrontal Cortex - Glutamate
Description: Glutamate brain metabolite levels between those with and without a lifetime history of prior alcohol abuse/dependence in the Left Dorsal Lateral Prefrontal Cortex (L DLPFC) using Magnetic Resonance Spectroscopy (MRS). Metabolite concentration was calculated from the MRS signals and reported in "mM".
Time Frame: Baseline screening (Scan 1) and again after 2 weeks of Acamprosate treatment (Scan 2)
Population: Usable scan data.
Measure: Mean (Standard Deviation); unit: mM
Arm/Group | ETOH Abuse | No ETOH Abuse
Number analyzed (Participants) | 13 | 14
mM
  Scan 1 | 7.45 (1.21) | 6.98 (1.07)
  Scan 2: number analyzed (Participants) | 11 | 12
  Scan 2 | 6.86 (1.03) | 6.92 (0.55)
  Difference: number analyzed (Participants) | 9 | 12
  Difference | -0.50 (1.36) | 0.03 (1.32)

14. Primary Outcome: Left Dorsal Lateral Prefrontal Cortex - N-acetylaspartate
Description: N-acetylaspartate (NAA) brain metabolite levels between those with and without a lifetime history of prior alcohol abuse/dependence in the Left Dorsal Lateral Prefrontal Cortex (L DLPFC) using Magnetic Resonance Spectroscopy (MRS). Metabolite concentration was calculated from the MRS signals and reported in "mM".
Time Frame: Baseline screening (Scan 1) and again after 2 weeks of Acamprosate treatment (Scan 2)
Population: Usable scan data.
Measure: Mean (Standard Deviation); unit: mM
Arm/Group | ETOH Abuse | No ETOH Abuse
Number analyzed (Participants) | 16 | 14
mM
  Scan 1 | 7.22 (0.99) | 7.50 (0.87)
  Scan 2: number analyzed (Participants) | 12 | 13
  Scan 2 | 7.44 (1.25) | 8.04 (1.68)
  Difference: number analyzed (Participants) | 12 | 12
  Difference | 0.25 (0.77) | 0.16 (0.91)

15. Primary Outcome: Left Dorsal Lateral Prefrontal Cortex - Myo-inositol
Description: Myo-inositol brain metabolite levels between those with and without a lifetime history of prior alcohol abuse/dependence in the Left Dorsal Lateral Prefrontal Cortex (L DLPFC) using Magnetic Resonance Spectroscopy (MRS). Metabolite concentration was calculated from the MRS signals and reported in "mM".
Time Frame: Baseline screening (Scan 1) and again after 2 weeks of Acamprosate treatment (Scan 2)
Population: Usable scan data.
Measure: Mean (Standard Deviation); unit: mM
Arm/Group | ETOH Abuse | No ETOH Abuse
Number analyzed (Participants) | 15 | 14
mM
  Scan 1 | 3.69 (0.79) | 3.61 (0.69)
  Scan 2: number analyzed (Participants) | 11 | 12
  Scan 2 | 3.34 (0.64) | 4.08 (0.91)
  Difference: number analyzed (Participants) | 10 | 12
  Difference | -0.08 (0.97) | 0.51 (0.72)

16. Primary Outcome: Fractional Anisotropy Measured With Diffusion Tensor Imaging
Description: Diffusion Tensor Imaging Frational Anisotropy (FA) Measures by Lifetime History of Alcohol Abuse/Dependence and Brain Hemisphere.
Time Frame: Completion of two scans
Population: Subjects completing study (both scans).
Measure: Mean (Standard Deviation); unit: FA
Arm/Group | ETOH Abuse | No ETOH Abuse
Number analyzed (Participants) | 13 | 15
FA
  Right hemisphere | 0.63 (0.03) | 0.61 (0.05)
  Left hemisphere | 0.59 (0.04) | 0.57 (0.04)

17. Secondary Outcome: BPRS - Symptoms of Psychosis Change in Scores
Description: Symptoms of psychosis were measured with the Brief Psychiatric Rating Scale (BPRS). The items rated for psychosis are "Conceptual Disorganization", "Suspiciousness", "Hallucinatory Behavior", and "Unusual Thought Content". Each item score ranges from "1=Not Present" to "7=Very Severe".
  Value at End of Study minus value at Baseline.
Time Frame: Baseline (Treatment Week 0) and End of Study (Treatment Week 2)
Population: Subjects completing the BPRS rating at Baseline and End of Study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ETOH Abuse | No ETOH Abuse
Number analyzed (Participants) | 11 | 16
units on a scale
  Conceptual Disorganization Change | -0.182 (0.603) | 0.0 (0.730)
  Suspiciousness Change | -0.636 (2.111) | -0.532 (1.209)
  Hallucinations Change | -0.0909 (1.7581) | -0.6250 (1.3102)
  Unusual Thought Content Change | -0.0909 (1.1362) | -0.1250 (0.7188)

18. Secondary Outcome: BPRS - Symptoms of Psychosis Total Score
Description: The psychosis total score is calculated by adding the scores for scales #4 Conceptual Disorganization, #11 Suspiciousness, #12 Hallucinatory Behavior, and #15 Unusual Thought Content. Each scale ranges from "1=Not Present" to "7=Very Severe". The minimum psychosis score is 4 and the maximum psychosis score is 28. A higher score indicates a more severe psychosis rating.
Time Frame: Baseline (Treatment Week 0) and End of Study (Treatment Week 2)
Population: Subjects completing BPRS rating at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ETOH Abuse | No ETOH Abuse
Number analyzed (Participants) | 16 | 17
units on a scale
  Baseline | 8.88 (3.77) | 9.47 (4.45)
  End of study: number analyzed (Participants) | 11 | 16
  End of study | 8.82 (4.14) | 8.38 (4.16)
  Change: number analyzed (Participants) | 11 | 16
  Change | -1.00 (3.95) | -1.31 (2.33)

19. Secondary Outcome: SANS - Negative Symptoms of Schizophrenia Total Score
Description: Negative symptoms of schizophrenia measured using the Scale for the Assessment of Negative Symptoms (SANS) Total Score. SANS total score range = 0-85. Higher scores indicate more severe negative symptoms.
Time Frame: Baseline (Treatment Week 0) and End of Study (Treatment Week 2)
Population: Subjects completing the SANS assessment at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ETOH Abuse | No ETOH Abuse
Number analyzed (Participants) | 16 | 17
units on a scale
  Baseline | 23.50 (10.73) | 26.12 (9.14)
  End of study: number analyzed (Participants) | 11 | 16
  End of study | 24.18 (12.09) | 26.38 (9.49)
  Change: number analyzed (Participants) | 11 | 16
  Change | 2.091 (8.384) | -0.375 (6.407)

20. Secondary Outcome: Cognitive Impairment
Description: Cognitive tests will include the DigitSymbol Test (evaluating processing speed), California Verbal Learning Test (CVLT; evaluating verbal learning and episodic memory), and NBack (evaluating working memory).
  Digit Symbol scaled scores range from 1 to 19, with the larger numbers indicating better performance.
  On the CVLT, the delayed recognition score ranges from 0 to 16, with the larger numbers indicating better performance.
  On the NBack test, subjects were asked to recall items 0-back, 1-back, and 2-back in a sequence. D-prime scores range from 0 to 8.6. Higher scores are better. As memory load increases from 0 to 1, from 1 to 2, D-prime scores are expected to be lower.
Time Frame: Change from Baseline (Treatment Week 0) to End of Study (Treatment Week 2)
Population: Subjects who completed cognitive testing at both study time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ETOH Abuse | No ETOH Abuse
Number analyzed (Participants) | 11 | 14
units on a scale
  Change in NBack 0-Back Total Hits | 0.000 (1.886) | 0.214 (1.188)
  Change in NBack 1-Back Total Hits | 0.60 (3.20) | 1.14 (3.42)
  Change in NBack 2-Back Total Hits | 1.70 (2.41) | 1.71 (3.27)
  Change in DigitSymbol Scaled Score | -0.20 (1.03) | 0.00 (1.30)
  Change in CVLT Total Recall | -0.600 (1.955) | -0.143 (1.956)

ADVERSE EVENTS:
Time Frame: Overall study of 6 weeks.
Description: Reportable adverse events (AEs) are defined as any harm experienced by a study participant, which in the opinion of the investigator is unexpected and probably related to the research procedures. None of our AEs met these criteria.
  Participants are systematically monitored for any increases the Side Effects Checklist (SEC). An SEC AE includes any symptom/side effect rated with a score of 4 (severe) or for which there was a 2 point change in severity from baseline.
Arm/Group | Single Arm
Serious Adverse Events (participants affected / at risk) | 0/36
Other Adverse Events (participants affected / at risk) | 6/36
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm (N=36)
Perceived increase in essential tremor (Nervous system disorders) | 1 (1) — Subject had a perceived increase in their essential tremor that they attributed to the study medication. Subject refused to continue participation.
Claustrophobia in MRI scan (Psychiatric disorders) | 1 (1) — Subject became claustrophobic in the MRI scanner. Refused to continue participation.
Diarrhea (Gastrointestinal disorders) | 3 (3)
Insomnia (General disorders) | 1 (1)
Restlessness (General disorders) | 1 (1)
Stiffness (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No